CLINICAL TRIAL: NCT03013361
Title: Comparison Ropivacaine and Bupivacaine in Sphenopalatine Ganglion Block for Postoperative Analgesia After Functional Endoscopic Sinus Surgery: A Randomized Controlled Trial
Brief Title: Ropivacaine and Bupivacaine in Sphenopalatine Ganglion Block in Sinus Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Sameer Sethi, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9157/PG2Trg/2012/15727
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Functional Endoscopic Sinus Surgery (FESS)
Keywords: ropivacaine, bupivacaine
MeSH Terms: interventions — Bupivacaine; Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group B (n=20) (Active Comparator): Group B (n=20): The patients in this group were infiltrated with 3 mL of 0.5% bupivacaine.
  Interventions: Drug: Bupivacaine
- Group R (n=20): (Active Comparator): Group R (n=20): The patients in this group were infiltrated with 3 mL of 0.5% ropivacaine.
  Interventions: Drug: Ropivacaine
- Group S (n=20, Control): (Placebo Comparator): Group S (n=20, Control): The patients in this group were infiltrated with 3 mL of normal saline.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Post operative pain control
  Other Names: Anawin
  Arms: Group B (n=20)
Drug: Ropivacaine — Post operative pain control
  Other Names: Ropin
  Arms: Group R (n=20):
Other: Normal Saline — Acts as comparator
  Other Names: Saline
  Arms: Group S (n=20, Control):

SUMMARY:
Postoperative analgesia after FESS can be achieved through opioids, NSAIDs, topical or infiltration of local anaesthetic and regional techniques like sphenopalatine ganglion (SPG) block, infraorbital nerve block and nasociliary block. As the current evidences regarding the benefit of SPG block after FESS is controversial, efficacy of sphenopalatine ganglion block will be evaluated using bupivacaine or ropivacaine as local anaesthetic in adult patients undergoing FESS under general anaesthesia in this study.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a minimally invasive and safe technique for the treatment of sinonasal disease. Although it is a minimally invasive and less traumatic procedure, it is usually associated with pain of mild to moderate intensity which reaches its maximum level in the first few postoperative hours. However, even low-level postoperative pain may be associated with delayed functional recovery and it frequently contributes to dissatisfaction with the procedure delay in return to work and readmission after surgery. Postoperative analgesia after FESS can be achieved through opioids, NSAIDs, topical or infiltration of local anaesthetic and regional techniques like sphenopalatine ganglion (SPG) block, infraorbital nerve block and nasociliary block. As the sensory innervations of the SPG supplies the nasal turbinates, nasopharynx and palate, SPG block is expected to provide perioperative analgesia after FESS. Integration of regional anaesthesia with general anaesthesia technique can provide a better hemodynamic control, less perioperative opioid use, less bleeding and higher level of patients' satisfaction. Reduction in surgical bleeding in FESS can improve surgical field and also surgeons' satisfaction and a reduced opioid use may be translated into a less postoperative nausea & vomiting, rapid recovery and early hospital discharge. But, the current evidences regarding the benefit of SPG block after FESS is controversial. In this randomized controlled trial, efficacy of sphenopalatine ganglion block will be evaluated using bupivacaine or ropivacaine as local anaesthetic in adult patients undergoing FESS under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 60 American Society of Anesthesiologists (ASA) physical status I and II patients
* aged 18-60 years scheduled to undergo elective functional endoscopic sinus surgery for sinonasal disease such as rhinosinusitis, polyps and deviated nasal septum were enrolled

Exclusion Criteria:

* Severe cardiovascular, pulmonary, hepatic, renal, neurologic or metabolic disease or coagulopathy
* History of allergy to any of the medications being used in the study
* Previous surgery for sinonasal disease
* Pre-existing chronic pain not related to chronic rhinosinusitis
* Taking prescription pain medications or antidepressants
* Chronic alcohol or drug abuse
* Inability to comprehend the study protocol
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary aim of the study was to assess the change in visual analogue scale comparing the effect of bilateral sphenopalatine ganglion block with bupivacaine and ropivacaine for postoperative analgesia after functional endoscopic sinus surgery | 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours thereafter.

SECONDARY OUTCOMES:
Time to first administration of rescue analgesia was recorded. | 8 hours
Patient satisfaction score | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Sethi, MD, Principal Investigator — PGIMER, Chandigarh,India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Ali A, Sakr S, Rahman A. Bilateral sphenopalatine ganglion block as adjuvant to general anaesthesia during endoscopic trans-nasal resection of pituitary adenoma. Egypt J Anaesth 2010;26;273-280. 2. Friedman M, Venkatesan TK, Lang D, Caldarelli DD. Bupivacaine for postoperative analgesia following endoscopic sinus surgery. Laryngoscope 1996;106:1382-1385. 3. Bicer C, Eskıtascıoglu T, Aksu R, Ulgey A, Yildiz K, Madenoglu H. Comparison of Preincisional Infiltrated Levobupivacaine and Ropivacaine for Acute Postoperative Pain Relief After Septorhinoplasty. Curr Ther Res Clin Exp 2011;72:13-22. 4. Fernandes SV. Postoperative care in functional endoscopic sinus surgery. Laryngoscope 1999;109:945-948.